CLINICAL TRIAL: NCT01945749
Title: Combined Intra Articular Corticosteroid and Physiotherapeutic Exercise in Patients With Osteoarthritis of the Knee: A Random-ised Clinical Trial
Brief Title: Exercise and Steroid in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101.04; 2012-002607-18 (EudraCT Number)
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intraarticular steroid + Exercise (Experimental): Intra-articular corticosteroid treatment with subsequent exercise therapy. Exercise therapy is commenced 2 weeks after injection
  Interventions: Drug: Intraarticular steroid; Other: Exercise therapy
- Intraarticular saline+Exercise (Active Comparator): Combined intra-articular saline injection and subsequent exercise therapy. Exercise therapy is commenced 2 weeks after injection
  Interventions: Drug: Intraarticular saline; Other: Exercise therapy

INTERVENTIONS:
Drug: Intraarticular steroid — 1 ml methylprednisolon corticosteroid (40 mg Depo-Medrol®) mixed with 4 ml Lidocain (10 mg/ml) without adrenalin. Injections are done ultrasound guided.
  Arms: Intraarticular steroid + Exercise
Drug: Intraarticular saline — 1 ml isotonic saline mixed with 4 ml Lidocain (10 mg/ml) without adrenalin. Injections are done ultrasound guided
  Arms: Intraarticular saline+Exercise
Other: Exercise therapy — The exercise is commenced 2 weeks after injection.
  The exercise includes a 10 minute warm up phase (ergometer bicycling) followed by strengthening and coordination exercises focusing on trunk, hip and knees.
  In case of pain or symptom exacerbation, a rescue exercise program is administered, excluding weight bearing activities.

SUMMARY:
Osteoarthritis (OA) of the knee is a very common chronic joint disorder associated pain and disability. As no cure exists, management aims to reduce pain, improve function, and enhance quality of life. The recommended hierarchy of management should consist of exercise in first line, then the add-on of drugs if necessary, and ultimately, if necessary, surgery.

The effect size of exercise therapy is of the same magnitude as most pharmacological treatments but is often without adverse effects. Local pharmacological treatment of the afflicted knee joint is recommended by means of intra-articular injections of corticosteroids, which is considered as a standard medical treatment of knee OA and are included in established guidelines for management of knee OA. While the two treatment approaches have been investigated separately in numerous clinical trials, the efficacy of a combined pharmacological and non-pharmacological approach is not known, despite the high rank of such combined treatment approach on the recommended hierarchy of management.

The purpose of this study is to assess the effects of exercise therapy in combination with intra-articular corticosteroid injections on patient reported pain and function in patients with knee OA.

The hypothesis is that the combined treatment approach (exercise therapy preceded by intra-articular injection of corticosteroid) enhances the clinical outcome compared to exercise therapy preceded by a placebo injection.

ELIGIBILITY:
Inclusion Criteria:

* age 40 years or above
* clinical knee osteoarthritis verified by radiography
* pain during level walking of at least 40 mm on a 0-100 mm visual analog scale
* clinical signs of local inflammation
* body mass index between 20 and 35

Exclusion Criteria:

* Exercise therapy within 3 months
* Intraarticular corticosteroid within 3 months
* Counter indications to exercise
* Counter indications to corticosteroid
* pregnant or breast feeding
* Auto immune disease
* Planned surgery in the study period
* significant cardiovascular disease
* significant neuroloigal disease
* significant psychiatric disease
* regional pain syndromes (e.g. fibromyalgia)
* spinal nerve root compression syndromes

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Knee pain | Change from baseline to week 14
  Self-reported pain assessed by the pain subdomain in the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire

SECONDARY OUTCOMES:
Knee pain | Change from baseline to week 2 and week 26
  Self-reported pain assessed by the pain subdomain in the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire
Knee symptoms | Change from baseline to week 2, 14, and 26
  Self-reported knee symptoms, knee related function, quality of life and, function during sports and recreation assessed by the pain subdomain in the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire
Functional pain test | Change from baseline to week 14, and 26
  Knee OA pain is associated with movement of the afflicted knee. Therefore we assess pain intensity and movement tolerance during repeated squatting. The test has 3 outcomes: 1) The number of pain free squatting movements that can be done in 30 seconds; 2) the number of painful squatting movements that can be done in 30 seconds; and 3) the average pain intensity during the squatting movements assessed on a 0-10 numeric rating scale.
Knee Muscle strength | Change from baseline to week 14, and 26
  Assessed by an isokinetic dynamometer
6 minute walk distance | Change from baseline to week 14, and 26
  The distance covered during 6 minutes of fast walking
Systemic markers of inflammation in blood | Change from baseline to week 14, and 26
  Blood sample
MRI based inflammation | Change from baseline to week 14, and 26
  To assess the severity and extent of local inflammation in the knee and surrounding tissues magnetic resonance imaging (MRI) are done before and after intravenous injection of a Gadolinium contrast agent. Contrast agents are only administered to participants with normal kidney function assessed from a standard blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Marius Henriksen, PhD, Study Chair — Frederiksberg University Hospital
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Dall CH, Andersen H, Povlsen TM, Henriksen M. Evaluation of a technology assisted physical activity intervention among hospitalised patients: A randomised study. Eur J Intern Med. 2019 Nov;69:50-56. doi: 10.1016/j.ejim.2019.08.019. Epub 2019 Sep 4. PMID 31494019
- [Derived] Bartholdy C, Klokker L, Bandak E, Bliddal H, Henriksen M. A Standardized "Rescue" Exercise Program for Symptomatic Flare-up of Knee Osteoarthritis: Description and Safety Considerations. J Orthop Sports Phys Ther. 2016 Nov;46(11):942-946. doi: 10.2519/jospt.2016.6908. Epub 2016 Sep 28. PMID 27681448
- [Derived] Henriksen M, Christensen R, Klokker L, Bartholdy C, Bandak E, Ellegaard K, Boesen MP, Riis RG, Bartels EM, Bliddal H. Evaluation of the benefit of corticosteroid injection before exercise therapy in patients with osteoarthritis of the knee: a randomized clinical trial. JAMA Intern Med. 2015 Jun;175(6):923-30. doi: 10.1001/jamainternmed.2015.0461. PMID 25822572